CLINICAL TRIAL: NCT00793780
Title: Pilot Trial of Naltrexone for Obesity in Women With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ethel F. Donaghue Women's Health Investigator Program at Yale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0808004106
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Schizophrenia; Schizoaffective Disorder
Keywords: obesity; schizophrenia; schizoaffective disorder; weight loss
MeSH Terms: conditions — Obesity; Schizophrenia; Psychotic Disorders; Weight Loss | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone 25mg (Active Comparator)
  Interventions: Drug: Naltrexone 25mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone 25mg — Naltrexone 25mg caplets taken orally once a day for 8 weeks
  Arms: Naltrexone 25mg
Other: Placebo — Placebo caplet (inactive substance) taken orally once a day for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to find out how effective low dose oral naltrexone is on reducing body weight when compared to placebo in women with schizophrenia and schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 to 70
* Meet DSM-IV (Diagnostic and Statistical Manual version IV) criteria for schizophrenia or schizoaffective disorder based on SCID (Structured Clinical Interview for the DSM-IV) interview
* Overweight, as defined with a BMI of equal to or greater than 27 kg/m² and continuing weight gain in the past year above 2% of previous years total body weight
* Be on a stable dose of antipsychotic medication; i.e. at least one month with no dosage change, and two months from an antipsychotic switch; 5) Deemed to be symptomatically stable by the clinical staff in the last two months

Exclusion Criteria:

* Meet criteria for current alcohol or other substance dependence, opioid use for any reason or positive urine drug screen for opiates
* A history of dementia, mental retardation or other neurological disorder that may interfere with study ratings
* Not capable of giving informed consent for participation in this study
* Ongoing pregnancy
* Known sensitivity to naltrexone
* A medical disorder that is known to cause obesity
* Use of sibutramine, topiramate, amphetamines or over the counter weight remedies
* Impaired liver functions (greater than 3 times the upper limit of normal)
* Diagnosed with polycystic ovary syndrome
* Currently being treated with insulin
* Current use of Depo-Provera or any natural/synthetic hormone treatment known to cause significant weight gain

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Result] Tek C, Ratliff J, Reutenauer E, Ganguli R, O'Malley SS. A randomized, double-blind, placebo-controlled pilot study of naltrexone to counteract antipsychotic-associated weight gain: proof of concept. J Clin Psychopharmacol. 2014 Oct;34(5):608-12. doi: 10.1097/JCP.0000000000000192. PMID 25102328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone 25mg | Placebo
Started | 12 | 12
Randomization | 12 | 12
Collected Baseline Data | 11 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Overweight women between the ages of 18 and 70 years who met the DSM-IV criteria for schizophrenia or schizoaffective disorder, on the basis of Structured Clinical Interview for DSM-IV. An additional participant dropped out of the study after baseline data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone 25mg | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9.6) | 41.4 (11.6) | 46.93 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 7 | 11
  Black | 7 | 4 | 11
  Hispanic | 0 | 1 | 1
Diagnosis [Number; unit: participants]
  Schizophrenia | 7 | 5 | 12
  Schizoaffective | 4 | 7 | 11
PANSS Total Score [Mean (Standard Deviation); unit: units on a scale] — The PANSS or the Positive and Negative Syndrome Scale is a medical scale used for measuring symptom severity of patients with schizophrenia. The scores for these scales are arrived at by summation of ratings across component items. Total score ranges from a minimum of 30 to a maximum of 210. A higher score indicates more severe symptoms.
  units on a scale | 64.7 (17.2) | 56.0 (16.7) | 59.78 (16.42)
Diabetes [Number; unit: participants]
  Diabetic | 6 | 1 | 7
  Non-Diabetic | 5 | 11 | 16
Years of education [Mean (Standard Deviation); unit: years] | 13.4 (4.1) | 13.7 (3.9) | 13.52 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From Baseline
Description: Weight was measured with shoes off to the nearest 0.1 kg.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
kg | -3.40 [-5.16 to -1.65] | 1.37 [-0.30 to 3.03]

2. Secondary Outcome: Fasting Serum Glucose Lab Values
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
mg/dL
  baseline | 113.40 (28.2) | 93.82 (7.9)
  Week 8 | 129.22 (45.2) | 94.11 (7.5)

3. Secondary Outcome: PANSS- Positive and Negative Symptom Scale
Description: The PANSS or the Positive and Negative Syndrome Scale is a medical scale used for measuring symptom severity of patients with schizophrenia. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale.The scores for these scales are arrived at by summation of ratings across component items. Total score ranges from a minimum of 30 to a maximum of 210. A higher score indicates more severe symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale | 57.50 (16.17) | 52.63 (17.91)

4. Secondary Outcome: Insulin Levels
Description: Determined with a double-antibody radioimmunoassay
Time Frame: baseline and week 8
Measure: Mean (Standard Deviation); unit: microIU/mL
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
microIU/mL
  baseline | 26.42 (40.0) | 13.84 (10.8)
  Week 8 | 35.51 (42.0) | 12.36 (4.4)

5. Secondary Outcome: LDL Cholesterol
Description: Determined by standard enzymatic procedures
Time Frame: baseline and week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
mg/dL
  baseline | 86.80 (26.2) | 123.18 (41.3)
  Week 8 | 104.11 (39.9) | 111.22 (33.5)

6. Secondary Outcome: Change in Questionnaire on Craving for Sweet or Rich Foods Score
Description: The Questionnaire on Craving for Sweet or Rich Foods (QCSRF) is a 2-factor, 9-item scale assessing the presence of cravings for rich and sweet foods and has been found to have good psychometric properties. The total score is the total of 2 sub scales. Total range is from 9 to 63, with a higher score indicative of a higher craving and reinforcement from sweet and/or rich foods.
Time Frame: baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone 25mg | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale | -3.10 (3.92) | 0 (4.31)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the start of medication, week 2, week 4, week 6 and week 8
Arm/Group | Naltrexone 25mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 9/10 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone 25mg (N=10) | Placebo (N=11)
Concentration (Psychiatric disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Sedation (General disorders) | 4 | 0
Failing Memory (Psychiatric disorders) | 1 | 0
Tension (General disorders) | 1 | 2
Increased Sleep (General disorders) | 3 | 0
Decreased Sleep (General disorders) | 1 | 0
Increased Dreaming (General disorders) | 1 | 2
Emotional Indifference (Psychiatric disorders) | 1 | 0
Dystonia (Musculoskeletal and connective tissue disorders) | 1 | 0
Rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tremor (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (General disorders) | 0 | 1
Increased Saliva (General disorders) | 1 | 0
Dry Mouth (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dizziness (General disorders) | 1 | 0
Photosensitivity (General disorders) | 2 | 0
Weight Loss (General disorders) | 3 | 1
Decreased Sexual Desire (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes